CLINICAL TRIAL: NCT00575536
Title: Optical Stimulation in Peripheral Nerves in Selective Rhizotomy Cases
Brief Title: Optical Stimulation in Peripheral Nerves for Select Rhizotomy Procedures
Acronym: Rhizotomy
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Anita Mahadevan-Jansen, Professor Biomedical Engineering and Neurosurgery, Vanderbilt University
Other Study IDs: 050822
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Spasticity
Keywords: spasticity; rhizotomy; surgery
MeSH Terms: conditions — Muscle Spasticity | interventions — Rhizotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — abnormal spinal nerves that have been surgically removed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Rhizotomy for children with spasticity: Children with spasticity needing Rhizotomy surgery
  Interventions: Procedure: Rhizotomy for children with spasticity

INTERVENTIONS:
Procedure: Rhizotomy for children with spasticity — Optical Stimulation versus electrical stimulation in children who need Rhizotomy Surgery for spasticity

SUMMARY:
The purpose of this study is to determine the safe and effective levels of optical stimulation in peripheral nerves of humans otherwise undergoing nerve lesioning in surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safe and effective levels of optical stimulation in peripheral nerves of humans otherwise undergoing nerve lesioning in surgery, namely children undergoing selective rhizotomy for treatment of medically refractory spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Children over the age of 3 and younger than 17 years
* Children who have failed appropriate medical therapy and are recommended for selective rhizotomy to treat spasticity by the pediatric neurosurgeon
* Children who would normally undergo electrodiagnostic testing including EMG monitoring for physiologic testing during surgery
* Surgery must be performed at the Vanderbilt University Children's Hospital

Exclusion Criteria:

* Patients in which a segment of the nerve (up to 2cm) cannot likely be identified at the time of surgery as determined by the pediatric neurosurgeon
* Children not undergoing routine selective rhizotomy for medically refractory spasticity as determined by the pediatric neurosurgeon
* Children who are medically unstable to tolerate an additional 20 minutes of experimental testing during the surgery
* Women who are pregnant will be excluded from this study

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children over the age of 3 and younger than 17 years who have failed appropriate medical therapy for spasticity and are recommended for Rhizotomy surgery
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
A brief series of optical versus electrical stimulation of the nerve will be used to measure the efficacy of optical stimulation | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Konrad, MD, Ph.D., Study Chair — Vanderbilt University, Dept. Neurosurgery; Chanqing Kao, MD, Ph.D., Principal Investigator — Vanderbilt University, Dept. Neurosurgery; Michael Remple, Ph.D., Principal Investigator — Vanderbilt University, Dept. Neurosurgery
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cayce JM, Wells JD, Malphrus JD, Kao C, Thomsen S, Tulipan NB, Konrad PE, Jansen ED, Mahadevan-Jansen A. Infrared neural stimulation of human spinal nerve roots in vivo. Neurophotonics. 2015 Jan;2(1):015007. doi: 10.1117/1.NPh.2.1.015007. Epub 2015 Feb 23. PMID 26157986